CLINICAL TRIAL: NCT00684450
Title: Cardiac Surgery : In Vivo Titration of Protamine
Brief Title: Cardiac Surgery: In Vivo Titration of Protamine
Acronym: Protamine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Organon (Industry)
Responsible Party: Principal Investigator, Antoine Rochon, M.D. FRCPC, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICM 07-997
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Bleeding
Keywords: titration of protamine; exact dose; protamine; neutralize heparin
MeSH Terms: conditions — Hemorrhage | interventions — Protamines; Cardiac Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): in vivo protamine titration in cardiac surgery. The titration is done during administration of protamine each 3 minutes to reach 2 consecutive ACT defined as 2 similar ACT values, within 10% variability, and ACT ≤ to 160 seconds. .The protamine is stopped when this values are obtain. Follow-up is done 15 minutes and 3 hours post-protamine
  Interventions: Procedure: Titration protamine
- 2 (Active Comparator): standard protamine administration ACT is done during administration of protamine each 3 minutes the values are recorded but the totality of protamine is given. Follow-up is done 15 minutes and 3 hours post-protamine
  Interventions: Drug: Standard administration of protamine

INTERVENTIONS:
Procedure: Titration protamine — 10. Study group: celite ACT will be performed every 3 minutes during protamine infusion until ACT values suggest reach of a plateau (defined as 2 similar ACT values, within 10% variability, and ACT ≤ to 160 seconds.), time at which infusion will be stopped. 2cc of blood is required per ACT test, for a maximum total of 10cc.
  Other Names: Protamine in vivo titration in cardiac surgery
  Arms: 1
Drug: Standard administration of protamine — 1.3 mg of Protamine for 100u héparine
  Arms: 2

SUMMARY:
Safe use of cardiopulmonary bypass (CPB) requires massive doses of intravenous unfractionated heparin. At end-CPB, residual heparin is neutralized with intravenous injection of protamine sulfate. This prospective, randomized, controlled study will be conducted in 82 voluntary subjects admitted for elective, first intention, cardiac surgery requiring cardiopulmonary bypass. Each will be randomly assigned to one of two groups. The control group will be submitted to a standard protamine infusion of 1.3mg :100U of the total heparin dose given during bypass. The test group will receive an infusion of protamine (over 15 minutes) until activated clotting time (ACT) values (determined every 3 minutes) depict a plateau, sign that the optimal protamine to heparin ratio has been attained. The investigators hypothesize this new in vivo titration method to be as efficient as the standard protocol (adequacy of heparin neutralization, % heparin rebound, bleeding, and transfusion), and potentially safer by its ability to prevent protamine overdose and its deleterious impact on platelet function.15

Principal Objective

Evaluate a new in vivo method of titration of protamine sulfate.

Secondary Objective

Evaluate the impact of this method on the adequacy of heparin neutralization by measuring:

1. platelet count
2. postoperative bleeding
3. transfusion exposure a
4. incidence of heparin rebound

DETAILED DESCRIPTION:
Protamine sulfate is administered to reverse the anticoagulant effects of heparin upon completion of cardiopulmonary bypass (CPB). In most cases, protamine is given in amounts sufficient to neutralize the total dose of heparin.9 This dose is usually calculated with a ratio of 1.3mg protamine for every 100U heparin given.10 In the literature, reported doses of intraoperatively administered protamine range from 0 to 8mg per 100U of heparin. Given in excess, protamine can, in addition to complement activation and hemodynamic instability,11 induce platelet dysfunctions.12-16 The latter significantly increases both the cost and morbidity of cardiac interventions as it is one of the main causes of postoperative bleeding. The optimal protamine/heparin ratio is difficult to individualize for each patient because of the great interpatient variability in heparin's metabolism4-7 and of the absence of correlation between ACT and heparin's plasma concentration.8 Consumption of heparin may vary from 0.01 to 3.86U/Kg per minute during CPB.30 The exact concentration of remaining circulating heparin at the end of bypass is not easily obtained.

ELIGIBILITY:
Inclusion Criteria:

* First intention, elective, cardiac surgery: either Coronary Artery Bypass Graft (CABG)or valve repair/replacement.
* Patients on preoperative aspirin, clopidogrel or heparin will be included.

Exclusion Criteria:

* Combination of CABG and valve surgery
* Second intention cardiac surgery
* ASA 5 patients
* Pre-existing hemostatic disorder (as evidenced by history)
* Pregnancy
* PLavix < 5 days before de surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Effective heparin neutralization (anti-Xa < 0.3 U/ml) | Pre protamine, 15 min post protamine, 3h post protamine

SECONDARY OUTCOMES:
Frequency of heparin rebound | 15 min post protamine and 3 hours post Protamine
Blood losses after surgery and transfusion requirements | discharge
Preservation of the platelet count | Pre operate, Pré Protamine, 15 min post Protamine, 3 hours post Protamine

CONTACTS AND LOCATIONS:
Overall Officials: Antoine G Rochon, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Hattersley PG. Activated coagulation time of whole blood. JAMA. 1966 May 2;196(5):436-40. No abstract available. PMID 5952227
- [Background] Young JA, Kisker CT, Doty DB. Adequate anticoagulation during cardiopulmonary bypass determined by activated clotting time and the appearance of fibrin monomer. Ann Thorac Surg. 1978 Sep;26(3):231-40. doi: 10.1016/s0003-4975(10)63676-4. PMID 110273
- [Background] Babka R, Colby C, El-Etr A, Pifarre R. Monitoring of intraoperative heparinization and blood loss following cardiopulmonary bypass surgery. J Thorac Cardiovasc Surg. 1977 May;73(5):780-2. PMID 850438
- [Background] McAvoy TJ. Pharmacokinetic modeling of heparin and its clinical implications. J Pharmacokinet Biopharm. 1979 Aug;7(4):331-54. doi: 10.1007/BF01062533. PMID 512841
- [Background] de Swart CA, Nijmeyer B, Roelofs JM, Sixma JJ. Kinetics of intravenously administered heparin in normal humans. Blood. 1982 Dec;60(6):1251-8. PMID 7139119
- [Background] Estes JW, Poulin PF. Pharmocokinetics of heparin. Distribution and elimination. Thromb Diath Haemorrh. 1975 Feb 28;33(1):26-37. No abstract available. PMID 47194
- [Background] Despotis GJ, Levine V, Joiner-Maier D, Joist JH. A comparison between continuous infusion versus standard bolus administration of heparin based on monitoring in cardiac surgery. Blood Coagul Fibrinolysis. 1997 Oct;8(7):419-30. doi: 10.1097/00001721-199710000-00007. PMID 9391723
- [Background] Gravlee GP, Case LD, Angert KC, Rogers AT, Miller GS. Variability of the activated coagulation time. Anesth Analg. 1988 May;67(5):469-72. No abstract available. PMID 3364767
- [Background] Despotis GJ, Gravlee G, Filos K, Levy J. Anticoagulation monitoring during cardiac surgery: a review of current and emerging techniques. Anesthesiology. 1999 Oct;91(4):1122-51. doi: 10.1097/00000542-199910000-00031. PMID 10519514
- [Background] Lowary LR, Smith FA, Coyne E, Dunham NW. Comparative neutralization of lung- and mucosal-derived heparin by protamine sulfate using in vitro and in vivo methods. J Pharm Sci. 1971 Apr;60(4):638-40. doi: 10.1002/jps.2600600436. No abstract available. PMID 5128383
- [Background] Kirklin JK, Chenoweth DE, Naftel DC, Blackstone EH, Kirklin JW, Bitran DD, Curd JG, Reves JG, Samuelson PN. Effects of protamine administration after cardiopulmonary bypass on complement, blood elements, and the hemodynamic state. Ann Thorac Surg. 1986 Feb;41(2):193-9. doi: 10.1016/s0003-4975(10)62668-9. PMID 3947172
- [Background] Carr ME Jr, Carr SL. At high heparin concentrations, protamine concentrations which reverse heparin anticoagulant effects are insufficient to reverse heparin anti-platelet effects. Thromb Res. 1994 Sep 15;75(6):617-30. doi: 10.1016/0049-3848(94)90174-0. PMID 7831681
- [Background] Harker LA. Bleeding after cardiopulmonary bypass. N Engl J Med. 1986 May 29;314(22):1446-8. doi: 10.1056/NEJM198605293142209. No abstract available. PMID 3702953
- [Background] Miyashita T, Nakajima T, Hayashi Y, Kuro M. Hemostatic effects of low-dose protamine following cardiopulmonary bypass. Am J Hematol. 2000 Jun;64(2):112-5. doi: 10.1002/(sici)1096-8652(200006)64:23.0.co;2-n. PMID 10814990
- [Background] Mochizuki T, Olson PJ, Szlam F, Ramsay JG, Levy JH. Protamine reversal of heparin affects platelet aggregation and activated clotting time after cardiopulmonary bypass. Anesth Analg. 1998 Oct;87(4):781-5. doi: 10.1097/00000539-199810000-00008. PMID 9768770
- [Background] Shigeta O, Kojima H, Hiramatsu Y, Jikuya T, Terada Y, Atsumi N, Sakakibara Y, Nagasawa T, Mitsui T. Low-dose protamine based on heparin-protamine titration method reduces platelet dysfunction after cardiopulmonary bypass. J Thorac Cardiovasc Surg. 1999 Aug;118(2):354-60. doi: 10.1016/S0022-5223(99)70227-8. PMID 10425010
- [Background] Berger RL, Ramaswamy K, Ryan TJ. Reduced protamine dosage for heparin neutralization in open-heart operations. Circulation. 1968 Apr;37(4 Suppl):II154-7. doi: 10.1161/01.cir.37.4s2.ii-154. No abstract available. PMID 5646575
- [Background] Guffin AV, Dunbar RW, Kaplan JA, Bland JW Jr. Successful use of a reduced dose of protamine after cardiopulmonary bypass. Anesth Analg. 1976 Jan-Feb;55(1):110-3. PMID 1108703
- [Background] Moriau M, Masure R, Hurlet A, Debeys C, Chalant C, Ponlot R, Jaumain P, Servaye-Kestens Y, Ravaux A, Louis A, Goenen M. Haemostasis disorders in open heart surgery with extracorporeal circulation. Importance of the platelet function and the heparin neutralization. Vox Sang. 1977;32(1):41-51. doi: 10.1111/j.1423-0410.1977.tb00602.x. PMID 841962
- [Background] Jobes DR, Schwartz AJ, Ellison N, Andrews R, Ruffini RA, Ruffini JJ. Monitoring heparin anticoagulation and its neutralization. Ann Thorac Surg. 1981 Feb;31(2):161-6. doi: 10.1016/s0003-4975(10)61536-6. PMID 6970019
- [Background] Ottesen S, Stormorken H, Hatteland K. The value of activated coagulation time in monitoring heparin therapy during extracorporeal circulation. Scand J Thorac Cardiovasc Surg. 1984;18(2):123-8. doi: 10.3109/14017438409102391. PMID 6611586
- [Background] Keeler JF, Shah MV, Hansbro SD. Protamine--the need to determine the dose. Comparison of a simple protamine titration method with an empirical dose regimen for reversal of heparinisation following cardiopulmonary bypass. Anaesthesia. 1991 Nov;46(11):925-8. doi: 10.1111/j.1365-2044.1991.tb09848.x. PMID 1750591
- [Background] Jobes DR, Aitken GL, Shaffer GW. Increased accuracy and precision of heparin and protamine dosing reduces blood loss and transfusion in patients undergoing primary cardiac operations. J Thorac Cardiovasc Surg. 1995 Jul;110(1):36-45. doi: 10.1016/S0022-5223(05)80007-8. PMID 7609566
- [Background] Shore-Lesserson L, Reich DL, DePerio M. Heparin and protamine titration do not improve haemostasis in cardiac surgical patients. Can J Anaesth. 1998 Jan;45(1):10-8. doi: 10.1007/BF03011985. PMID 9466020
- [Background] Despotis GJ, Joist JH, Hogue CW Jr, Alsoufiev A, Kater K, Goodnough LT, Santoro SA, Spitznagel E, Rosenblum M, Lappas DG. The impact of heparin concentration and activated clotting time monitoring on blood conservation. A prospective, randomized evaluation in patients undergoing cardiac operation. J Thorac Cardiovasc Surg. 1995 Jul;110(1):46-54. doi: 10.1016/S0022-5223(05)80008-X. PMID 7609568
- [Background] Hardy JF, Belisle S, Robitaille D, Perrault J, Roy M, Gagnon L. Measurement of heparin concentration in whole blood with the Hepcon/HMS device does not agree with laboratory determination of plasma heparin concentration using a chromogenic substrate for activated factor X. J Thorac Cardiovasc Surg. 1996 Jul;112(1):154-61. doi: 10.1016/s0022-5223(96)70191-5. PMID 8691862
- [Background] Gravlee GP, Rogers AT, Dudas LM, Taylor R, Roy RC, Case LD, Triscott M, Brown CW, Mark LJ, Cordell AR. Heparin management protocol for cardiopulmonary bypass influences postoperative heparin rebound but not bleeding. Anesthesiology. 1992 Mar;76(3):393-401. doi: 10.1097/00000542-199203000-00012. PMID 1539851
- [Background] Martin P, Horkay F, Gupta NK, Gebitekin C, Walker DR. Heparin rebound phenomenon--much ado about nothing? Blood Coagul Fibrinolysis. 1992 Apr;3(2):187-91. PMID 1606290
- [Background] Shanberge JN, Murato M, Quattrociocchi-Longe T, van Neste L. Heparin-protamine complexes in the production of heparin rebound and other complications of extracorporeal bypass procedures. Am J Clin Pathol. 1987 Feb;87(2):210-7. doi: 10.1093/ajcp/87.2.210. PMID 3812352
- [Background] Mabry CD, Read RC, Thompson BW, Williams GD, White HJ. Identification of heparin resistance during cardiac and vascular surgery. Arch Surg. 1979 Feb;114(2):129-34. doi: 10.1001/archsurg.1979.01370260019002. PMID 426618